CLINICAL TRIAL: NCT03664011
Title: A Phase I, Open-label, Single-dose Trial to Investigate Metabolism and Pharmacokinetics of BI 730357 BS (C-14) Administered as Oral Solution in Healthy Male Volunteers
Brief Title: A Study in Healthy Men to Test How BI 730357 is Processed by the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1407-0031; 2018-001837-41 (EudraCT Number)
Record Dates: First submitted 2018-09-07; First posted 2018-09-10 (Actual); Results first posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2022-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BI 730357 BS (C-14) (Experimental): All participants were administered an oral single dose of 50 milligram (mg) BI 730357 containing [C-14] BI 730357 base (BS) (pure 14C-labelled "hot" drug substance) and BI 730357 BS (unlabelled "cold" drug substance). This mixture corresponds to the warm substance BI 730357 BS (C-14) containing a radioactive dose of approximately 3.7 MegaBecquerel (MBq), (100 microcurie (µCi)), and was administered in a solution of 10 milliliter (mL) volume with 240 mL of water after an overnight fast of at least 10 hours (h).
  Interventions: Drug: BI 730357 mixed with [C-14]BI 730357 BS

INTERVENTIONS:
Drug: BI 730357 mixed with [C-14]BI 730357 BS — Oral Solution

SUMMARY:
The main objectives of the study are as follows:

* To assess the mass balance recovery of (C-14) BI 730357-radioactivity (also expressed as 14C-BI 730357-EQ) in urine and faeces after a single oral dose of 50 mg BI 730357 base (BS) (C-14) in healthy male subjects
* To provide plasma, urine, and faecal samples for metabolite profiling and structural identification

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 65 years (incl.)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with good clinical practice (GCP) and local legislation
* Subjects who are sexually active must use, with their partner, highly effective contraception from the time of administration of trial medication until 4 months after administration of trial medication. Adequate methods are:

  * Condoms plus use of hormonal contraception by the female partner that started at least 2 months prior to administration of trial medication (e.g. implants, injectables, combined oral or vaginal contraceptives, intrauterine device) or
  * Condoms plus surgical sterilization (vasectomy at least 1 year prior to enrolment) or
  * Condoms plus surgically sterilised partner (including hysterectomy) or
  * Condoms plus intrauterine device or
  * Condoms plus partner of non-childbearing potential (including homosexual men) Subjects are required to use condoms to prevent unintended exposure of the partner to the study drug via seminal fluid. Male and female condoms must not be used together. Alternatively, true abstinence is acceptable when it is in line with the subjec's preferred and usual lifestyle. If a subject is usually not sexually active but becomes active, with their partner, they must comply with the contraceptive requirements detailed above.

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 139 mmHg, diastolic blood pressure outside the range of 45 to 89 mmHg, or pulse rate outside the range of 40 to 100 bpm.
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Clinically significant gastrointestinal (including known or suspected inflammatory bowel disease), hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* Further exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PRA Health Sciences Onderzoekscentrum Martini, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https:// www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was planned to include healthy male participants in this non-randomised, open-label, single-arm, single-dose trial. They were recruited from the volunteer's pool of the study site.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI 730357: All participants were administered an oral single dose of 50 milligram (mg) BI 730357 containing [C-14] BI 730357 base (BS) (pure 14C-labelled "hot" drug substance) and BI 730357 BS (unlabelled "cold" drug substance). This mixture corresponds to the warm substance BI 730357 BS (C-14) containing a radioactive dose of approximately 3.7 MegaBecquerel (MBq), (100 microcurie (µCi)), and was administered in a solution of 10 milliliter (mL) volume with 240 mL of water after an overnight fast of at least 10 hours (h).
Period: Overall Study
Arm/Group | BI 730357
Started (Started are treated) | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS) :This subject set included all participants who were documented to have received one dose of trial medication.
Arm/Group | BI 730357
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.2 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mass Balance Recovery of Total [14C]-Radioactivity in Urine (Feurine, 0-tz)
Description: feurine, fractions of [14C]-radioactivity excreted in urine as percentage of the administered dose over the time interval from 0 to tz, where tz is the latest quantifiable data point across all participants.
Time Frame: Within 18 hours (h) predose, 0-4, 4-8, 8-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168, 168-192, 192-216, 216-240, 240-264, 264-288, 288-312, 312-336 h after dosing on Day 1, continued in 24 h intervals, every 7 days from Day 21 until Day 50.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): The PKS included all subjects in the TS who provided at least one value for primary or secondary PK endpoints and were not excluded due to relevant protocol deviations or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of administered dose (%)
Arm/Group | BI 730357
Number analyzed (Participants) | 6
Percentage of administered dose (%) | 34.3 (19.2)

2. Primary Outcome: Mass Balance Recovery of Total [14C]-Radioactivity in Faeces (Fefaeces, 0-tz)
Description: fefaeces, 0-tz, fraction of [14C]-radioactivity excreted in faeces as percentage of the administered dose over the time interval from 0 to tz, where tz is the latest quantifiable data point across all participants.
Time Frame: Within 48 hours (h) predose, 0-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168, 168-192, 192-216, 216-240, 240-264, 264-288, 288-312 and 312-336 h after dosing on Day 1 and continued in 24 h intervals, every 7 days up to Day 50.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of administered dose (%)
Arm/Group | BI 730357
Number analyzed (Participants) | 6
Percentage of administered dose (%) | 65.0 (8.09)

3. Secondary Outcome: Maximum Measured Concentration of 14C-BI 730357-equivalent (EQ) and BI 730357 (Cmax)
Description: Cmax, maximum measured concentration of 14C-BI 730357-equivalent (EQ) and BI 730357 in plasma after a single oral dose of 50 mg BI 730357 BS (C-14) is presented. Plasma concentrations of (C-14) BI 730357-radioactivity are expressed as 14C-BI 730357-EQ.
Time Frame: Within 3:00 Hours: minutes (h:m) pre-dose, 0:30, 1:00, 1:30, 2:00, 4:00, 8:00, 12:00, 24:00, 48:00, 72:00, 120:00, 168:00, 216:00, 264:00, 312:00, 485:00, 653:00 and 821:00 after drug administration.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomole/litre (nmol/L)
Groups:
- 14C-BI 730357-EQ and BI 730357: All participants were administered an oral single dose of 50 milligram (mg) BI 730357 containing [C-14] BI 730357 base (BS) (pure 14C-labelled "hot" drug substance) and BI 730357 BS (unlabelled "cold" drug substance). This mixture corresponds to the warm substance BI 730357 BS (C-14) containing a radioactive dose of approximately 3.7 MegaBecquerel (MBq), (100 microcurie (µCi)), and was administered in a solution of 10 milliliter (mL) volume with 240 mL of water after an overnight fast of at least 10 hours (h).
Arm/Group | 14C-BI 730357-EQ and BI 730357
Number analyzed (Participants) | 6
Nanomole/litre (nmol/L)
  14C-BI 730357-EQ | 1020 (16.5)
  BI 730357 | 641 (19.2)

4. Secondary Outcome: Area Under the Concentration-time Curve of 14C-BI 730357-equivalent (EQ) and BI 730357 Over the Time Interval From 0 to the Last Quantifiable Time Point (AUC0-tz)
Description: AUC0-tz, area under the concentration-time curve of 14C-BI 730357-equivalent (EQ) and BI 730357 over the time interval from 0 to the last quantifiable time point in plasma after a single oral dose of 50 mg BI 730357 BS (C-14) is presented. Plasma concentrations of (C-14) BI 730357-radioactivity are expressed as 14C-BI 730357-EQ.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomole*Hours/litre (nmol*h/L)
Arm/Group | 14C-BI 730357-EQ and BI 730357
Number analyzed (Participants) | 6
Nanomole*Hours/litre (nmol*h/L)
  14C-BI 730357-EQ | 24300 (50.8)
  BI 730357 | 9410 (79.9)

ADVERSE EVENTS:
Time Frame: From drug administration until End-of-trial (EoT) examination, up to 50 days.
Arm/Group | BI 730357
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 730357 (N=6)
Catheter site haematoma (General disorders) | 1
Catheter site inflammation (General disorders) | 1
Vessel puncture site haematoma (General disorders) | 1
Headache (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT03664011/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT03664011/SAP_001.pdf